CLINICAL TRIAL: NCT03161990
Title: Debridement, Antibiotics and Implant Retention (DAIR) for Infected Total Hip Arthroplasty- Does the Operative Approach Influence the Functional Result?
Brief Title: DAIR for Infected Total Hip Arthroplasty - Does the Operative Approach Influence the Functional Result?
Status: Completed | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Asbjorn Aroen, Professor, University Hospital, Akershus
Other Study IDs: 287901
Record Dates: First submitted 2017-05-15; First posted 2017-05-22 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Hip Prosthesis Infection; Arthroplasty Complications
Keywords: DAIR; Transgluteal approach; Posterior approach

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transgluteal approach to the hip joint: Patients who have been revised once for an infected total hip replacement with debridement and implant retention and in whom both the primary hip arthroplasty and the revision procedure were performed through a transgluteal approach.
  Interventions: Procedure: Transgluteal approach to the hip joint
- Posterior approach to the hip joint: Patients who have been revised once for an infected total hip replacement with debridement and implant retention and in whom both the primary hip arthroplasty and the revision procedure were performed through a posterior approach.
  Interventions: Procedure: Posterior approach to the hip joint

INTERVENTIONS:
Procedure: Transgluteal approach to the hip joint — Operative approach to the hip joint where the abductors are partly detached from the greater trochanter and the hip joint is approached through the anterior part of the capsule.
  Other Names: Direct lateral approach to the hip joint
  Groups: Transgluteal approach to the hip joint
Procedure: Posterior approach to the hip joint — Operative approach to the hip joint where the short external rotators are detached from the greater trochanter and the hip joint is approached through the posterior part of the capsule.
  Other Names: Posterolateral approach to the hip joint
  Groups: Posterior approach to the hip joint

SUMMARY:
The functional outcome and quality of life after treatment for an infected hip arthroplasty have been found to be significantly worse compared to an uncomplicated arthroplasty. However, the type of revision surgery chosen to treat the infection plays a role for the functional outcome. The concept of DAIR (debridement, antibiotics and implant retention) has been shown to yield god results with respect to infection control in cases of early infection with a stable implant and better functional results than a to-stage revision. In patients where infection control was achieved after just one DAIR procedure the functional outcome was comparable to an uncomplicated primary arthroplasty. However, it is not known if the operative approach used for the primary and revision surgery plays a role for the functional result after treatment of an infected total hip arthroplasty with DAIR. The project's aim is to investigate if the choice of the operative approach (transgluteal or posterior) for the primary hip replacement and the revision surgery has an influence on the functional result after debridement and implant retention for an infected total hip replacement.

DETAILED DESCRIPTION:
Potential study participants will be identified in the Norwegian Arthroplasty Register. Patients who have been revised once for an infected total hip arthroplasty with debridement and implant retention and in whom either the transgluteal og posterior operative approach was used in both procedures will be selected. The potential participants will be contacted by letter. They will be asked for written informed consent and to fill out three questionnaires: the Hip Disability Osteoarthritis Score (HOOS), which also allows for the calculation of the Western Ontario and McMaster Universities osteoarthritis index (WOMAC), the EQ-5D (quality of life) and a questionnaire asking about confirmation that the patient only has been revised once for his/her infected arthroplasty, about limping, other complications (nerve injury, dislocation, reoperation for other causes than infection), if the infection is considered to have been eradicated and overall satisfaction. The data recorded in the Norwegian Arthroplasty Register will be used in a multiple linear regression analysis to evaluate if the surgical approach is an independent factor influencing the outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* The infected total hip arthroplasty has only been revised once.
* The revision procedure was a debridement and implant retention.
* Both, the primary and the revision procedure were performed through the same surgical approach; either the transgluteal or the posterior approach.

Exclusion Criteria:

* No written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The potential study participant will be identified in the Norwegian Arthroplasty Register.
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2018-11-17 (Actual); Study Completion 2018-11-17 (Actual)

PRIMARY OUTCOMES:
Function subscale score of the WOMAC | At minimum 1 year, on average 5 year follow-up from the DAIR procedure
  Function subscale score of the Western Ontario and McMaster Universities osteoarthritis index (WOMAC)

SECONDARY OUTCOMES:
WOMAC score | At minimum 1 year, on average 5 year follow-up from the DAIR procedure
  Western Ontario and McMaster Universities osteoarthritis index score
HOOS | At minimum 1 year, on average 5 year follow-up from the DAIR procedure
  Hip Disability Osteoarthritis Score
EQ-5D score | At minimum 1 year, on average 5 year follow-up from the DAIR procedure
  Quality of life score
Limping | At minimum 1 year, on average 5 year follow-up from the DAIR procedure
  Patient reported limping on the side of the revised total hip replacement.
Other complications | At minimum 1 year, on average 5 year follow-up from the DAIR procedure
  Patient reported nerve injury, dislocation, reoperation for other causes than infection.
Overall satisfaction | At minimum 1 year, on average 5 year follow-up from the DAIR procedure
  Overall satisfaction with the revised total hip replacement assessed by questionnaire.

OTHER OUTCOMES:
Infection eradication | At minimum 1 year, on average 5 year follow-up from the DAIR procedure
  Patient reported eradication of the infection of their total hip arthroplasty.

CONTACTS AND LOCATIONS:
Overall Officials: Asbjorn Aaroen, Professor, Study Director — University Hospital, Akershus
Locations (1):
- Akershus University hospital, Lørenskog, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cahill JL, Shadbolt B, Scarvell JM, Smith PN. Quality of life after infection in total joint replacement. J Orthop Surg (Hong Kong). 2008 Apr;16(1):58-65. doi: 10.1177/230949900801600115. PMID 18453662
- [Background] Byren I, Bejon P, Atkins BL, Angus B, Masters S, McLardy-Smith P, Gundle R, Berendt A. One hundred and twelve infected arthroplasties treated with 'DAIR' (debridement, antibiotics and implant retention): antibiotic duration and outcome. J Antimicrob Chemother. 2009 Jun;63(6):1264-71. doi: 10.1093/jac/dkp107. Epub 2009 Mar 31. PMID 19336454
- [Background] Grammatopoulos G, Kendrick B, McNally M, Athanasou NA, Atkins B, McLardy-Smith P, Taylor A, Gundle R. Outcome Following Debridement, Antibiotics, and Implant Retention in Hip Periprosthetic Joint Infection-An 18-Year Experience. J Arthroplasty. 2017 Jul;32(7):2248-2255. doi: 10.1016/j.arth.2017.02.066. Epub 2017 Mar 6. PMID 28385345
- [Derived] Pollmann CT, Gjertsen JE, Dale H, Straume-Naesheim TM, Dybvik E, Hallan G. Operative approach influences functional outcome after DAIR for infected total hip arthroplasty. Bone Joint J. 2020 Dec;102-B(12):1662-1669. doi: 10.1302/0301-620X.102B12.BJJ-2020-0501.R1. PMID 33249901